CLINICAL TRIAL: NCT04704297
Title: Trigger Point Injection for Myofascial Pain Syndrome in the Low Back (T-PIMPS): A Randomized Controlled Trial.
Brief Title: Trigger Point Injection for Myofascial Pain Syndrome in the Low Back: A Randomized Controlled Trial
Acronym: T-PIMPS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joshua Oliver, Emergency Medicine Physician / Assistant Research Director Department of Emergency Medicine, Madigan Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 220042
Record Dates: First submitted 2020-12-28; First posted 2021-01-11 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Low Back Pain; Myofascial Pain Syndrome Lower Back
Keywords: Trigger Point Injection; Low Back Pain; Myofascial Pain Syndrome; Emergency Department
MeSH Terms: conditions — Low Back Pain; Myofascial Pain Syndromes; Emergencies | interventions — Ketorolac; Acetaminophen; Ibuprofen; cyclobenzaprine; Bupivacaine; Saline Solution; Aftercare

STUDY DESIGN:
Intervention Model Description: This will be a prospective three-armed randomized controlled trial. There will be no crossover. The first arm will be single blinded as it will be obvious to the investigators that it does not involve trigger point injections. The other two arms will be double blinded trigger point injections with either Bupivacaine or Normal Saline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The two trigger point injection arms will be drawn-up and randomized by a research pharmacist prior to delivery to the Emergency Department. These two army will be Bupivacaine and Normal Saline, which are identical in appearence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Standard Therapy (ST) (Active Comparator): ST will consist of 975mg of Acetaminophen PO and either 30mg of Ketorolac IM or 15 mg IV. Upon discharge ST will consist of prescriptions for acetaminophen 650mg every 4 hours by mouth, Ibuprofen 400mg every 4 hours by mouth, and 10 mg of cyclobenzaprine nightly by mouth. Additionally, participants will be provided a handout going over these medications and the use of heat for low back pain and instructions on the performance of McKenzie stretching exercises for low back pain.4
  Interventions: Drug: Treatment of Myofascial Pain Syndrome in the low back. This intervention will be based on outcomes of the medications listed below.; Drug: Evaluation of functional ability using a patient centered functional score known as the Modified Oswestry Disability Index (MODI). The intervention will be based on outcomes of medications below.; Drug: Following up with participants 60-72 hours after treatment in the Emergency Department. This intervention will be based on outcomes of the medications listed below.
- ST plus Trigger Point Injections (TPI) with 8 mL of 0.5 percent Bupivacaine (Active Comparator): ST plus TPI with 8 mL of 0.5 percent Bupivacaine
  Interventions: Drug: Treatment of Myofascial Pain Syndrome in the low back. This intervention will be based on outcomes of the medications listed below.; Drug: Evaluation of functional ability using a patient centered functional score known as the Modified Oswestry Disability Index (MODI). The intervention will be based on outcomes of medications below.; Drug: Following up with participants 60-72 hours after treatment in the Emergency Department. This intervention will be based on outcomes of the medications listed below.
- ST plus TPI with 8 mL of Normal Saline (NS) (Active Comparator): ST plus TPI with 8 mL of Normal Saline
  Interventions: Drug: Treatment of Myofascial Pain Syndrome in the low back. This intervention will be based on outcomes of the medications listed below.; Drug: Evaluation of functional ability using a patient centered functional score known as the Modified Oswestry Disability Index (MODI). The intervention will be based on outcomes of medications below.; Drug: Following up with participants 60-72 hours after treatment in the Emergency Department. This intervention will be based on outcomes of the medications listed below.

INTERVENTIONS:
Drug: Treatment of Myofascial Pain Syndrome in the low back. This intervention will be based on outcomes of the medications listed below. — We are testing which of the three arms is superior for the treatment of Myofascial Pain Syndrome of the Low Back. Pain will be measured using a 10 cm visual analogue scale (VAS) at baseline and 30-minutes after treatment.
  Other Names: Ketorolac, acetaminophen, ibuprofen, cyclobenzaprine, bupivacaine, normal saline
Drug: Evaluation of functional ability using a patient centered functional score known as the Modified Oswestry Disability Index (MODI). The intervention will be based on outcomes of medications below. — Evaluation of functional ability using a patient centered functional score known as the MODI. The MODI will be scored at baseline and 30-minutes after treatment.
  Other Names: Ketorolac, acetaminophen, ibuprofen, cyclobenzaprine, bupivacaine, normal saline
Drug: Following up with participants 60-72 hours after treatment in the Emergency Department. This intervention will be based on outcomes of the medications listed below. — 60-72 after treatment in the Emergency Department, a member of the study team will follow up with participants to repeat a measurement of pain and functional ability on VAS and MODI respectively. This will be compared to baseline measurements.
  Other Names: Ketorolac, acetaminophen, ibuprofen, cyclobenzaprine, bupivacaine, normal saline

SUMMARY:
Rationale: Low back pain (LBP), or myofascial pain syndrome (MPS) of the low back, accounts for approximately 2.63 million visits in the United States, or 2.3 percent of annual Emergency Department (ED) visits. An estimated 100 billion dollars per year is lost from LBP. Approximately one-third of this is direct costs. Previous studies have established the safety of trigger point injections (TPI). However, the results of these studies are highly heterogeneous regarding TPI's ability to treat pain or improve functional outcomes. The two most promising TPI studies conducted in the ED have been published in the last two years. They both suffered from a small sample size. Additionally, they suffered from a combination of limitations including: lack of randomization, inconsistent medical management, lack of a follow-up assessment, and lack of patient centered functional outcomes. These studies were both two armed and either compared standard medical management to TPI with local anesthetic or TPI with local anesthetic to TPI with Normal Saline (NS). One of these studies concluded that TPI is generally beneficial. The other concluded that TPI with NS is superior.

Research Hypothesis: The investigators hypothesize that standard therapy (ST) plus TPI with 8 mL of 0.5 percent Bupivacaine is superior to ST alone or ST plus TPI with 8 mL of NS for the treatment of the pain associated with MPS of the low back.

Significance: This will be the first TPI study to compare ST, to TPI with local anesthetic, and TPI with NS for LBP conducted in an ED. It will also be the first TPI study to incorporate a patient centered functional outcome and patient follow-up after discharge from an ED. TPI's are a popular treatment modality for LBP among many Emergency Medicine Providers. However, to date, there is limited evidence for or against it. The investigators are hopeful that this study will answer whether or not trigger point injections are benefiting patients and, if so, which type of TPI is most beneficial.

DETAILED DESCRIPTION:
Significance: Low back pain (LBP) is a common presenting complaint in the Emergency Department (ED), accounting for 2.63 million visits in the united states and 2.3 percent of ED visits annually.1 An estimated 100 billion dollars per year is lost from low back pain. One-third of this is direct costs.2 For the United States military, in 2015, 195,844 acute cases of LBP were identified, leading to significant loss of person-hours.3 The definitions of durations, or types, of LBP vary among sources. For example, the American Association of Family Physicians defines acute low back pain as six to 12 weeks of pain and chronic pain as anything more than 12 weeks.4 A more specific definition used by The American College of Physicians defines acute LBP from 0-4 weeks, subacute LBP as 5-12 weeks, and chronic low back pain as greater than 12 weeks.5 A specific definition of chronic low back pain is essential if including acute on chronic low back pain in a study. These specific definitions will not only be used for demographics, they will also aid in excluding other causes of LBP from the study such as fibromyalgia, rheumatoid arthritis, and ankylosing spondylitis.6,7 The investigators will include exacerbations of chronic LBP, but they will have to satisfy a specific definition. An excepted definition of an exacerbation of chronic low back pain is an increase of 1.5 cm above baseline pain on a 10 cm visual analog scale (VAS). The justification is that this is outside the standard deviation of typical back pain estimations.8 As this study of LBP focuses on TPIs, the investigators are narrowing the definition of LBP to myofascial pain syndrome (MPS) of the low back. The investigators chose this definition as MPS is defined by trigger points.9 Use of MPS is also consistent with prior TPI studies of LBP.10-15 The trigger points of MPS are recognized clinically by having two out of three of the following criteria: a taut band of muscle on exam, reproduction of pain upon palpation, and referred pain along a band of muscle upon palpation.16-18 The two most promising TPI studies previously conducted in the ED have been published in the last two years.19,20 They both suffered from a small sample size. Additionally, they suffered from a combination of limitations including: lack of randomization, inconsistent medical management, lack of a follow-up assessment, and lack of patient centered functional outcomes.19,20 These studies were both two armed and either compared standard medical management to TPI with local anesthetic or TPI with local anesthetic to TPI with Normal Saline (NS).19,20 One of these studies concluded that TPIs are generally beneficial.19 The other concluded that TPIs with NS are superior.20 The investigators endeavor to complete a randomized controlled trial (RCT) that definitively answers whether TPIs with local anesthetic are superior to TPIs with NS in an ED setting. The investigators will also be comparing both of these treatments to standard therapy (ST). Bupivacaine was chosen as it is the longest acting commonly available local anesthetic in most EDs.21 The investigators hypothesize that TPIs with Bupivacaine are superior to TPIs with NS or ST. If the investigators are correct this simple and inexpensive treatment could have a large impact on the financial burden and loss in person-hours caused by MPS of the low back.1-3,21

Innovation:

The invistigators will innovate by building upon lessons learned from previous TPI studies for MPS conducted in the ED.19,20 The study has also been designed with the best practices of CONSORT standards in mind.22 Unlike previous studies, this RCT will include three groups, ST, ST plus TPI with Bupivacaine, and ST plus TPI with NS. Additionally, each of these treatment arms will be highly regimented to improve the quality of evidence the investigators produce. The investigators will also follow up with study participants via telephone at 60-72 hours to determine if the treatment provided more than temporary pain relief. Lastly, the investigators will incorporate a patient centered functional score.23 A measure of functional ability is particularly relevant to MPS given its associated cost in lost person-hours.2 To date, such an endeavor to investigate TPIs in the ED has not been undertaken.

Approach:

This study will be conducted in the Emergency Department at Madigan Army Medical Center on Joint Base Lewis-McChord in Tacoma, WA. This is an academic center and level II trauma center with an annual Emergency Department census of 60,000. It is home to an Emergency Medicine Residency program and serves as a tertiary referral center for Department of Defense personnel in the Pacific Region. This study has approval from the local Institutional Review Board.

This study is a prospective 3-armed RCT. The first arm will be ST. The second army will be ST plus TPI with 8 mL of 0.5 percent Bupivacaine. The third arm will be ST plus TPI with 8 mL of NS. The first arm will be single blinded as it will be obvious to medical professionals that the patient is not receiving trigger points. The remaining two arms will be double blinded. The ST arm will be highly standardized to eliminate variation in treatment. It will also contain no narcotics or benzodiazepines. ST will consist of 975mg of Acetaminophen PO and either 30mg of Ketorolac IM or 15 mg IV. Upon discharge ST will consist of prescriptions for acetaminophen 650mg every 4 hours by mouth, Ibuprofen 400mg every 4 hours by mouth, and 10 mg of cyclobenzaprine nightly by mouth. If a potential participant is allergic to any of the study medications, they cannot participate. Additionally, participants will be provided a handout going over these medications and the use of heat for low back pain and instructions on the performance of McKenzie stretching exercises for low back pain.4 Bupivacaine was chosen as it is the longest acting local anesthetic commonly available in most EDs. With a toxic dose of 2mg/Kg, 8 mL is well within safety limits for the study population as it only contains 40mg of Bupivacaine.21 NS was chosen as the third arm as it is the primary TPI treatment that local anesthetic TPIs are compared to, Bupivacaine and NS are also identical in appearance.12,21 It is possible that participants will be able to tell which TPI they have received based on Bupivacaine's anesthetic properties.21 To address this, the investigators will be asking participants that received a TPI to guess which medication they received on the data collection form. 30-minutes following study medication administration, data will be collected. 60-72 hours after treatment is initiated, telephone follow-up will be completed by a member of the study team. This time frame was chosen as it is a clinically relevant timeframe for ED bounce backs.24 Additionally, this time frame is well beyond four half-lives of Bupivacaine (2.7 hours x 4 = 10.8 hours).21 This ensures that the data collected at telephone follow-up will not be influenced by any lingering impact of the medication.

The investigators plan to begin enrolling participants January 2nd, 2021. The institution's Research Pharmacist will contact one of the institution's statisticians to obtain a randomization scheme. The investigators will then be sent pre-drawn up and pre-randomized medications for storage in the ED medication refrigerator. Participants randomized to ST will be represented by empty syringes.

The investigators plan to enroll participants as a convenience sample. Although continuous enrollment would be ideal, the research team consists of nine investigators, five of which are Emergency Medicine Residents. Given off-service rotations and a small research team, providing 24-hour coverage for enrollment is not feasible. Review of the EDs census over the last three months revealed that the ED sees a minimum of 40 patients a month for the chief complaint (CC) of "low back pain". A review of the census in the three month prior to the COVID-19 outbreak revealed that this number is less than half of the number of patients the investigators usually see for the CC of "low back pain". This is very likely due to a decreased ED utilization rates for non-emergent CC's during COVID-19. The investigators suspect that as vaccinations become more widely available, these numbers will normalize. However, if the census remained as is and the investigators operate under the assumption that the investigators could reasonably capture 50 percent of the LBP patients that came through the Emergency Department, it would take us a minimum of nine months to complete the study. With these assumptions, enrollment would be complete in June of 2022.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Must have at least 1 trigger point in low back paraspinal muscles.
3. For exacerbations of chronic low back pain, the pain on presentation must be 1.5 cm above baseline pain on VAS

Exclusion Criteria:

1. Allergy or inability to take study medications.
2. New focal neurologic deficit in lower extremities.
3. Known active malignancy with bony spinal metastases.
4. Identifiable spinal, lumbosacral or hip fracture.
5. History of Fibromyalgia, rheumatoid arthritis, ankylosing spondylitis.
6. Current use of anticoagulation.
7. Overlying cellulitis.
8. Spinal, hip, or pelvic surgery within the past 6 months.
9. Previous administration of trigger point injections for current episode.
10. Sciatica-extending down the back of the leg to the heel.
11. Alternate identifiable cause of participant's acute pain other than myofascial or musculoskeletal pain.
12. Febrile patients.
13. Pregnant
14. Unable to understand English or otherwise unable to provide informed consent (mental handicap, inability to understand instructions, risks, or benefits), or is an at risk population (wounded warrior, resident physicians, prisoners, cadets, midshipmen, or students).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-12-28 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain reduction | 30-minutes
  To determine which of three treatments is the superior treatment for myofascial pain syndrome (MPS) of the low back. The three treatments are standard therapy (ST), ST plus trigger point injections (TPI) with 8 mL of 0.5% Bupivacaine, and ST plus TPI with 8 mL of normal saline NS. To reach superiority a treatment will have to decrease pain by 1.5 cm more than the other treatments, measured before treatment and 30-minutes following treatment on a 10 cm visual analog scale (VAS). The units of measurement are centimeters (cm) on a VAS.

SECONDARY OUTCOMES:
Functional Improvement | 30-minutes
  To incorporate a patient centered functional score into the study and measure the difference in scores before treatment and 30-minutes following treatment. We will use the Modified Oswestry Disability Index (MODI), a previously validated index. To reach superiority, a treatment will have to decrease MODI by 10 points more than the other treatments. The MODI produces a measurement in percentages ranging from 0 to 100. The measurement will therefore be a percentage.

OTHER OUTCOMES:
Follow-up measurement of pain | 60-72 hours
  To follow-up with participants via telephone 60-72 hours after treatment and repeat a pain measurement on a 10 cm VAS. The same measures of superiority will be applied comparing the baseline measurement to the measurement at 60-72 hours. The unit of measurement will be cm on a VAS.
Follow-up measurement of function | 60-72 hours
  To follow-up with participants via telephone 60-72 hours after treatment and repeat a functional score on a MODI. The same measures of superiority will be applied comparing the baseline measurement to the measurement at 60-72 hours. The unit of measurement will be percentage on a MODI.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua J Oliver, MD, Principal Investigator — Madigan AMC
Locations (1):
- Department of Emergency Medicine, Madigan Army Medical Center, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: No
We plan to report our data on clinical trials.gov, but we do not plan to share it.

REFERENCES:
- [Background] Friedman BW, Chilstrom M, Bijur PE, Gallagher EJ. Diagnostic testing and treatment of low back pain in United States emergency departments: a national perspective. Spine (Phila Pa 1976). 2010 Nov 15;35(24):E1406-11. doi: 10.1097/BRS.0b013e3181d952a5. PMID 21030902
- [Background] Luo X, Pietrobon R, Sun SX, Liu GG, Hey L. Estimates and patterns of direct health care expenditures among individuals with back pain in the United States. Spine (Phila Pa 1976). 2004 Jan 1;29(1):79-86. doi: 10.1097/01.BRS.0000105527.13866.0F. PMID 14699281
- [Background] Dietrich EJ, Leroux T, Santiago CF, Helgeson MD, Richard P, Koehlmoos TP. Assessing practice pattern differences in the treatment of acute low back pain in the United States Military Health System. BMC Health Serv Res. 2018 Sep 17;18(1):720. doi: 10.1186/s12913-018-3525-8. PMID 30223830
- [Background] Casazza BA. Diagnosis and treatment of acute low back pain. Am Fam Physician. 2012 Feb 15;85(4):343-50. PMID 22335313
- [Background] Chou R, Deyo R, Friedly J, Skelly A, Weimer M, Fu R, Dana T, Kraegel P, Griffin J, Grusing S. Systemic Pharmacologic Therapies for Low Back Pain: A Systematic Review for an American College of Physicians Clinical Practice Guideline. Ann Intern Med. 2017 Apr 4;166(7):480-492. doi: 10.7326/M16-2458. Epub 2017 Feb 14. PMID 28192790
- [Background] Harden RN, Bruehl SP, Gass S, Niemiec C, Barbick B. Signs and symptoms of the myofascial pain syndrome: a national survey of pain management providers. Clin J Pain. 2000 Mar;16(1):64-72. doi: 10.1097/00002508-200003000-00010. PMID 10741820
- [Background] Chandola HC, Chakraborty A. Fibromyalgia and myofascial pain syndrome-a dilemma. Indian J Anaesth. 2009 Oct;53(5):575-81. PMID 20640108
- [Background] Dernek B, Adiyeke L, Duymus TM, Gokcedag A, Kesiktas FN, Aksoy C. Efficacy of Trigger Point Injections in Patients with Lumbar Disc Hernia without Indication for Surgery. Asian Spine J. 2018 Apr;12(2):232-237. doi: 10.4184/asj.2018.12.2.232. Epub 2018 Apr 16. PMID 29713403
- [Background] Han SC, Harrison P. Myofascial pain syndrome and trigger-point management. Reg Anesth. 1997 Jan-Feb;22(1):89-101. doi: 10.1016/s1098-7339(06)80062-3. PMID 9010953
- [Background] Roldan CJ, Huh BK. Iliocostalis Thoracis-Lumborum Myofascial Pain: Reviewing a Subgroup of a Prospective, Randomized, Blinded Trial. A Challenging Diagnosis with Clinical Implications. Pain Physician. 2016 Jul;19(6):363-72. PMID 27454266
- [Background] Hong CZ. Lidocaine injection versus dry needling to myofascial trigger point. The importance of the local twitch response. Am J Phys Med Rehabil. 1994 Jul-Aug;73(4):256-63. doi: 10.1097/00002060-199407000-00006. PMID 8043247
- [Background] Frost FA, Jessen B, Siggaard-Andersen J. A control, double-blind comparison of mepivacaine injection versus saline injection for myofascial pain. Lancet. 1980 Mar 8;1(8167):499-500. doi: 10.1016/s0140-6736(80)92761-0. PMID 6102230
- [Background] Lugo LH, Garcia HI, Rogers HL, Plata JA. Treatment of myofascial pain syndrome with lidocaine injection and physical therapy, alone or in combination: a single blind, randomized, controlled clinical trial. BMC Musculoskelet Disord. 2016 Feb 24;17:101. doi: 10.1186/s12891-016-0949-3. PMID 26911981
- [Background] Ay S, Evcik D, Tur BS. Comparison of injection methods in myofascial pain syndrome: a randomized controlled trial. Clin Rheumatol. 2010 Jan;29(1):19-23. doi: 10.1007/s10067-009-1307-8. Epub 2009 Oct 20. PMID 19838864
- [Background] Raeissadat SA, Rayegani SM, Sadeghi F, Rahimi-Dehgolan S. Comparison of ozone and lidocaine injection efficacy vs dry needling in myofascial pain syndrome patients. J Pain Res. 2018 Jun 29;11:1273-1279. doi: 10.2147/JPR.S164629. eCollection 2018. PMID 29988746
- [Background] Alvarez DJ, Rockwell PG. Trigger points: diagnosis and management. Am Fam Physician. 2002 Feb 15;65(4):653-60. PMID 11871683
- [Background] Lavelle ED, Lavelle W, Smith HS. Myofascial trigger points. Anesthesiol Clin. 2007 Dec;25(4):841-51, vii-iii. doi: 10.1016/j.anclin.2007.07.003. PMID 18054148
- [Background] Shah JP, Thaker N, Heimur J, Aredo JV, Sikdar S, Gerber L. Myofascial Trigger Points Then and Now: A Historical and Scientific Perspective. PM R. 2015 Jul;7(7):746-761. doi: 10.1016/j.pmrj.2015.01.024. Epub 2015 Feb 24. PMID 25724849
- [Background] Yanuck J, Saadat S, Lee JB, Jen M, Chakravarthy B. Pragmatic Randomized Controlled Pilot Trial on Trigger Point Injections With 1% Lidocaine Versus Conventional Approaches for Myofascial Pain in the Emergency Department. J Emerg Med. 2020 Sep;59(3):364-370. doi: 10.1016/j.jemermed.2020.06.015. Epub 2020 Jul 22. PMID 32712034
- [Background] Roldan CJ, Osuagwu U, Cardenas-Turanzas M, Huh BK. Normal Saline Trigger Point Injections vs Conventional Active Drug Mix for Myofascial Pain Syndromes. Am J Emerg Med. 2020 Feb;38(2):311-316. doi: 10.1016/j.ajem.2019.158410. Epub 2019 Aug 24. PMID 31477359
- [Background] Shen JJ, Taylor DM, Knott JC, MacBean CE. Bupivacaine in the emergency department is underused: scope for improved patient care. Emerg Med J. 2007 Mar;24(3):189-93. doi: 10.1136/emj.2006.040253. PMID 17351224
- [Background] Hopewell S, Clarke M, Moher D, Wager E, Middleton P, Altman DG, Schulz KF; CONSORT Group. CONSORT for reporting randomized controlled trials in journal and conference abstracts: explanation and elaboration. PLoS Med. 2008 Jan 22;5(1):e20. doi: 10.1371/journal.pmed.0050020. PMID 18215107
- [Background] Vianin M. Psychometric properties and clinical usefulness of the Oswestry Disability Index. J Chiropr Med. 2008 Dec;7(4):161-3. doi: 10.1016/j.jcm.2008.07.001. PMID 19646379

DOCUMENTS (1):
  • Informed Consent Form (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT04704297/ICF_000.pdf